CLINICAL TRIAL: NCT01153139
Title: Long-term Bilateral Theta Burst Stimulation for the Treatment of Major Depression
Acronym: TheBuS_D
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Prof. Dr. med., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 124/2009BO1
Record Dates: First submitted 2010-04-23; First posted 2010-06-29 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Major Depression
Keywords: Transcranial Magnetic Stimulation; Depression; Theta Burst Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bilateral theta burst stimulation to the DLPFC (Experimental): intermittent TBS (iTBS) to the left DLPFC continuous TBS (cTBS) to the right DLPFC
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation, TBS)
- Sham stimulation (Placebo Comparator): Sham stimulation with a 45° tilted coil
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation, TBS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (Theta Burst Stimulation, TBS) — intermittent TBS (iTBS) to the left DLPFC (600 stimuli, 80% resting motor threshold) continuous TBS (cTBS) to the right DLPFC (600 stimuli, 80% resting motor threshold)

SUMMARY:
Repetitive transcranial magnetic stimulation has been shown to be moderately effective in the treatment of major depression. Theta burst stimulation (TBS) is a new form of rTMS that may exert larger effects.

This sham-controlled study examines the effectivity of daily bilateral TBS to the dorsolateral frontal cortex over 6 weeks in 2x16 patients with major depression add on to the local standard of a combined pharmacological/psychotherapeutical treatment.

ELIGIBILITY:
Inclusion Criteria:

* major Depression
* informed consent

Exclusion Criteria:

* seizures in medical history
* metallic implants
* deep brain stimulation
* cardiac pacemaker
* brain trauma
* psychotic symptoms
* substance abuse
* pregnancy
* Benzodiazepines other than Lorazepam >1mg/d

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of responders (response = decrease of the Montgomery-Åsberg Depression Rating Scale for at least 50%) | after the end of treatment (week 6)

SECONDARY OUTCOMES:
Change of the Hamilton rating scale for depression (HAMD 17) | baseline, after the end of treatment (week 6)
Change of the Beck Depression Inventory (BDI) | baseline, after the end of treatment (week 6)
Change of the Montgomery-Asberg rating scale for depression (MADRS) score | baseline, after the end of treatment (week 6)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tübingen, Department of Psychiatry and Psychotherapy, Tübingen, Germany